CLINICAL TRIAL: NCT02342769
Title: Prospective Non-Interventional Observational Study of Use of Triumeq® and Corresponding Monitoring Measures in Clinical Practice in Germany
Brief Title: Prospective Non-Interventional Observational Study of Use of TRIUMEQ and Corresponding Monitoring Measures in Clinical Practice in Germany
Acronym: TRIUMPH
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 202033
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dolutegravir/Abacavir/Lamivudin: Prospective, non-interventional observational study on the use of TRIUMEQ and the respective monitoring measures in the practice of HIV care in Germany. No drug will be provided. No study visits or procedures are mandated per protocol.
  Interventions: Drug: Dolutegravir/Abacavir/Lamivudin

INTERVENTIONS:
Drug: Dolutegravir/Abacavir/Lamivudin — Prospective, non-interventional observational study on the use of TRIUMEQ and the respective monitoring measures in the practice of HIV care in Germany. No drug will be provided. No study visits or procedures are mandated per protocol.

SUMMARY:
TRIUMPH is a prospective, non-interventional observational study on the use of the fixdose combination TRIUMEQ (Dolutegravir/Abacavir/Lamivudine) and the respective monitoring measures in the practice of HIV care in Germany. The primary study objective is a descriptive report of the incidence of therapeutic monitoring measures in HIV-infected patients under TRIUMEQ therapy in everyday routine practice in Germany. The study is designed to enroll approximately 400 patients. There are no protocol-mandated visits or procedures associated with the study. Each patient is expected to participate for a maximum of 3 years or until premature discontinuation (i.e., discontinuation of TRIUMEQ, due to death, withdrawal of consent, lost to follow-up. TRIUMEQ is a registered trademark of the ViiV Healthcare group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Age ≥ 18 years
* HLA-B*5701-negative
* Decision for first initiation of TRIUMEQ therapy made by the attending physician independent of the inclusion in this observational study

Exclusion Criteria:

* Prior dolutegravir therapy (cf. also Capping ABC in section 3.3 Recruitment)
* Participation in a clinical trial during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approx. 40 HIV treatment sites in Germany are planned to be involved in the documentation. The recruitment target is to include a total of 400 patients in the study across Germany. In order to allow for adequately answering in particular the problems regarding HLA-B*5701 testing, at least half of the recruited population should not have received abacavir (ABC) in their prior therapy. Each site will be allowed to recruit a maximum of 5 patients per month and a maximum of 20 patients in total. If the monthly quota of 5 patients is not utilized, the difference may be transferred to the subsequent months.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2018-10-28 (Actual)

PRIMARY OUTCOMES:
Frequency of therapeutic monitoring measures in HIV-infected patients | up to 3 years
  Descriptive documentation of the frequency of therapeutic monitoring measures in HIV-infected patients under TRIUMEQ in routine daily practice in Germany

SECONDARY OUTCOMES:
Type of the therapeutic monitoring measures | up to 3 years
  Descriptive characterization of therapeutic monitoring measures in HIV-infected patients under TRIUMEQ in routine daily practice in Germany
Details on conduct and logistics of HLA-B*5701 testing | Baseline
  Descriptive characterization of conduct and logistics of HLA-B*5701 testing in HIV-infected patients under TRIUMEQ in routine daily practice in Germany
Number of participants with Serious Adverse Events and drug-related adverse events as a measure of safety and tolerability | up to 3 years
  To evaluate the frequency and type of serious adverse events and drug-related adverse events in patients treated with dolutegravir
Efficacy | up to 3 years
  Defined as viral load < 50 copies/ml
Resistance profile | up to 3 years
  To characterise resistance profile in case of virological failure
Patient satisfaction | up to 3 years
  To evaluate the change in patient satisfaction relative to baseline in patients treated with TRIUMEQ
Reasons for selecting TRIUMEQ | Baseline
Reasons for discontinuing TRIUMEQ | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (18):
- Germany (18):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Chemnitz
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Dortmund
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Weimar